CLINICAL TRIAL: NCT01614652
Title: Percutaneous Ventricular Restoration in Chronic Heart Failure Due to Ischemic Heart Disease
Brief Title: A Pivotal Trial to Establish the Efficacy and Long-term Safety of the Parachute Implant System
Acronym: PARACHUTE IV
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company is closed
Sponsor: CardioKinetix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VA0956
Record Dates: First submitted 2012-06-04; First posted 2012-06-08 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Congestive Heart Failure; Left Ventricular (LV) Systolic Dysfunction
Keywords: Congestive Heart Failure Due to LV Systolic Dysfunction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parachute Implant and All Appropriate Medical Therapy (AAMT) (Experimental)
  Interventions: Device: CardioKinetix Parachute Implant and All Appropriate Medical Therapy (AAMT)
- All Appropriate Medical Therapy (AAMT) (No Intervention)

INTERVENTIONS:
Device: CardioKinetix Parachute Implant and All Appropriate Medical Therapy (AAMT) — CardioKinetix Parachute implant and all appropriate medical therapy
  Arms: Parachute Implant and All Appropriate Medical Therapy (AAMT)

SUMMARY:
Treatment of ischemic heart failure.

ELIGIBILITY:
Candidates for this study must meet ALL of the following inclusion criteria:

Clinical Inclusion Criteria:

* Age ≥ 18 and ≤ 79 years.
* Body Mass Index (BMI) ≤ 40.
* Symptomatic ischemic heart failure (New York Heart Association (NYHA) Class III or "ambulatory" Class IV as determined through the use of the SAS) post Myocardial Infarction (MI) in the Left Anterior Descending (LAD) territory at least 60 days prior to enrollment.
* Patient is not hospitalized at the time of enrollment.
* Receiving appropriate medical treatment for heart failure according to the current American College of Cardiology (ACC)/American Heart Association (AHA) Guideline Update for the Diagnosis and Management of Chronic Heart Failure in the Adult during the three months prior to enrollment.
* The patient or the patient's legal representative has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent as approved by the Institutional Review Board (IRB)/Ethics Committee (EC) of the respective clinical site.
* The patient and the treating physician agree that the patient will return for all required post-procedure follow-up visits.

Inclusion Criteria based on Imaging:

* 15% ≤ Left Ventricular Ejection Fraction (LVEF) ≤ 35% by Transthoracic Echocardiogram (TTE).
* Post LV MI structural heart dysfunction represented by LV wall motion abnormality (WMA) by TTE.
* Left ventricle must have appropriate anatomy (size and morphology) for implant placement using Cardiac Computed Tomography (CT) and confirmed by LV gram

Candidates will be excluded from the study if ANY of the following conditions apply:

Clinical Exclusion Criteria:

* Untreated clinically significant coronary artery disease requiring revascularization.
* Cardiogenic shock within 72 hours of enrollment.
* Patient has received a pacemaker, Implantable Cardioverter Defibrillator (ICD), or Cardiac Resynchronization Therapy (CRT) within 60 days of enrollment.
* Excessive wall motion abnormalities outside the anteroapical region.
* Recent (within 6 months) cerebrovascular accident (CVA) or transient ischemic attack (TIA).
* End stage renal disease requiring chronic dialysis.
* Obstructive Sleep Apnea (OSA): unless compliant on CPAP therapy or successful surgery.
* Hemoglobin < 10 g/dl (female), < 12 g/dl (male) or Creatinine > 2.5mg/dl.
* Blood dyscrasia, history of bleeding diathesis or coagulopathy, or hypercoagulable states.
* Active peptic ulcer or GI bleeding within the past 3 months.
* A known hypersensitivity or contraindication to aspirin, warfarin, nitinol (titanium and nickel alloy), or sensitivity to contrast media, which cannot be adequately pre-medicated.
* Ongoing sepsis, including active endocarditis.
* Life expectancy < 1 year due to associated non-cardiac co-morbid conditions or currently on the heart transplant lists.
* Other medical, social, or psychological conditions that in the opinion of an Investigator precludes the patient from appropriate consent.
* Currently participating in an investigational drug or another device study (prior to primary endpoint reached).
* Female patients with childbearing potential and a positive urine pregnancy test .

Anatomical Exclusion Criteria:

* Pre-existing prosthetic heart valve in mitral or aortic position.
* Valvular stenosis or regurgitation (tricuspid, aortic or mitral) > 2+.
* Presence of anatomic anomalies (including severe calcification) detected by cardiac imaging (echocardiogram, Computed Tomography (CT), or LV gram) preventing unimpeded deployment and/or operation of the Parachute Implant

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2012-12; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Death or re-hospitalization for Worsening Heart Failure (WHF) | At least 1 year

CONTACTS AND LOCATIONS:
Overall Officials: William T Abraham, MD, Principal Investigator — Ohio State University; Marco A Costa, MD, PhD, Principal Investigator — University Hospitals; Leslie Saxon, MD, Principal Investigator — University of Southern California
Locations (68):
- United States (67):
  - Arizona Heart, Phoenix, Arizona
  - University of Arizona Medical Center, Tucson, Arizona
  - Arkansas Heart, Little Rock, Arkansas
  - University of Southern California (USC), Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Morton Plant Hospital - Heart and Vascular Institute of Florida, Clearwater, Florida
  - Delray Medical Center, Delray Beach, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Florida Hospital Tampa - Pepin Heart Institute, Tampa, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Kootenai Heart Clinics, Coeur d'Alene, Idaho
  - Evanston Hospital, Evanston, Illinois
  - Advocate Medical Group - Midwest Heart Foundation, Naperville, Illinois
  - Prairie Education and Research Cooperative - St. John's Hospital, Springfield, Illinois
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Iowa Heart Center, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - St Joseph Hospital/Kentucky One, Lexington, Kentucky
  - Jewish Hospital/Louisville, Louisville, Kentucky
  - Cardiovascular Institute of the South, Houma, Louisiana
  - LSU Health Sciences Center, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - St. Joseph Mercy-Michigan Heart, Ann Arbor, Michigan
  - MidMichigan Medical Center, Midland, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - St. Luke's MAHI, Kansas City, Missouri
  - Nebraska Heart Hospital, Lincoln, Nebraska
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Hackensack UMC, Hackensack, New Jersey
  - Gates Vascular Institute/Buffalo General Hospital, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Univ. Of Rochester Medical Center, Rochester, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - The Christ Hospital Lindner Research Center, Cincinnati, Ohio
  - University Hospitals, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Ohio Health Research Institute/Riverside Methodist Hospital, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Einstein Healthcare Network Cardiology, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center - Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Wormleysburg, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Tennova Healthcare - Turkey Creek Medical Center, Knoxville, Tennessee
  - Saint Thomas West Hospital, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - Texas Heart Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Inova Heart and Vascular, Fairfax, Falls Church, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Costa MA, Pencina M, Nikolic S, Engels T, Templin B, Abraham WT. The PARACHUTE IV trial design and rationale: percutaneous ventricular restoration using the parachute device in patients with ischemic heart failure and dilated left ventricles. Am Heart J. 2013 Apr;165(4):531-6. doi: 10.1016/j.ahj.2012.12.022. Epub 2013 Feb 19. PMID 23537969